CLINICAL TRIAL: NCT02306941
Title: Internet-delivered Cognitive Behavior Therapy for Functional Abdominal Pain in Adolescents - an Open Pilot.
Brief Title: Internet-delivered CBT for Functional Abdominal Pain in Adolescents - a Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAP pilot ICBT 2015
Record Dates: First submitted 2014-11-30; First posted 2014-12-03 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Functional Gastrointestinal Disorders; Abdominal Pain; Dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases; Abdominal Pain; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-delivered CBT (Experimental): 10 sessions of ICBT during 10 weeks for the adolescents. 5 session of parent training during 10 weeks for parents. Therapist support is provided at least once weekly through the platform developed for the purpose. Therapists are trained CBT-psychologists.
  Interventions: Behavioral: Internet-delivered CBT

INTERVENTIONS:
Behavioral: Internet-delivered CBT — The Internet-delivered exposure treatment is based on the well-established internet-delivered CBT-treatment for IBS in adults, adapted for adolescents with FAP/FD and their parents. Main component in the treatment is exposure for symptoms. The purpose of the treatment is to reduce fearful and anxious responses to symptoms and lessen avoidance of symptoms in the adolescents, and to teach the parents how parental behavior can influence symptoms in children as well as how to support exposure. Detailed behaviour analysis is made for each individual and instruction is given on how to gradually expose to symptoms to lessen fear for symptoms and widen the behavioral repertoire.

SUMMARY:
This pilot-study aims to evaluate the treatment effects and feasibility of an internet-delivered CBT-program adjusted for adolescents with functional abdominal pain and functional dyspepsia.

DETAILED DESCRIPTION:
Functional abdominal pain (FAP) and functional dyspepsia, are common in adolescents and associated with impaired quality of life. In adults with IBS, internet-delivered CBT leads to reduced symptoms and increased quality of life, but studies in children are lacking. This pilot-study aim to evaluate the treatment effects and feasibility of an internet-delivered CBT-program for adolescents with FAP and FD.

Method: Pilot study with a pre-post-design and no control group. The internet-delivered CBT-program will last for 10 weeks and include weekly therapist support, consisting of online messages and telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 at inclusion date
* fulfilling Rome III-criteria for FAP or FD with:

  1. a written diagnosis from patient's physician and negative required tests (Blood samples: C-reactive protein or erythrocyte sedimentation rate, Blood count and IgA-Transglutaminase. Stool: f-Calprotectin)
  2. The Rome III questionnaire + clinical interview confirming the diagnosis

Exclusion Criteria:

* Concurrent serious medical conditions
* Concurrent serous psychiatric diagnosis
* On-going psychological treatment
* Absence from school exceeding an average of 2 days a week is a cause for exclusion since high absence demands more intensive interventions than can be offered in ICBT
* On-going abuse or severe parental psychiatric illness in the family
* Pronounced language skill deficits and learning difficulties lead to exclusion from the study
* Lack of regular internet-access

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Faces pain scale - R | Baseline to 12 weeks.
  Change in pain intensity measured with a self-rating scale daily during 2 weeks at baseline and daily during 10th to 12th week post treatment for analysis of effect.The Faces Pain Scale is a self-report measure used to assess the intensity of children's pain. Faces have four faces representing least pain and most pain on equal intervals on a scale from 0-10. Its validity is supported by a strong positive correlation (r=0.93, N=76) with a visual analogue scale (VAS) measure in children aged 5-12 years. The metric for scoring (0-10) conforms closely to a linear interval scale.

SECONDARY OUTCOMES:
Faces pain scale - R | Baseline to 9 months
  Change in pain intensity measured with a self-rating scale daily during 2 weeks at baseline and daily during 2 weeks after 9 months for analysis of effect.The Faces Pain Scale is a self-report measure used to assess the intensity of children's pain. Faces have four faces representing least pain and most pain on equal intervals on a scale from 0-10. Its validity is supported by a strong positive correlation (r=0.93, N=76) with a visual analogue scale (VAS) measure in children aged 5-12 years. The metric for scoring (0-10) conforms closely to a linear interval scale.
Faces pain scale - R | Weekly during treatment (treatment week 1-9).
  Change in pain intensity measured with a self-rating scale weekly during treatment for mediation analyses.
Gastrointestinal Symptom Rating Scale-IBS Version (GSRS-IBS) | Baseline to 10 weeks, baseline to 9 months
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 10 weeks, and from baseline to 9 months for analysis of effect.The GSRS-IBS have 13 items about weekly gastrointestinal symptoms like bloating, hard stool, abdominal pain etc. It is a seven-point Likert scale from 1 (no discomfort at all) to 7 (very severe discomfort). The GSRS-IBS has excellent psychometric properties with internal consistency between α = .74 (for abdominal pain) to α = .85 (for satiety).
IBS-behavioral responses questionnaire (IBS-BRQ) | Weekly during treatment (treatment week 1-9). Baseline to 10 weeks, baseline to 9 months.
  Change in Gastrintestinalsymptoms-specific behaviors measured with a self-rating scale weekly during treatment for mediation analyses, and from baseline to 10 weeks, baseline to 9 months, for analysis of effect. The scale consists of 26 items on a seven-point Likert scale from 1 (never) to 7 (always). The scale includes items related to avoidance behavior such as "I avoid certain social situations (e.g. restaurants) because of my symptoms " and to toilet behavior such as "I spend more time on the toilet than ideally I would like". IBS-BRQ is both reliable and valid with a high degree of internal consistency for adults with IBS (Cronbach's α=.86). The scale differentiate significantly between IBS patients and healthy controls (F=221, P<.01).
Percieved Stress scale (PSS 10) | Weekly during treatment (treatment week 1-9). Baseline to 10 weeks, baseline to 9 months.
  Change in perceived stress measured with a self-rating scale weekly during treatment for mediation analyses, and from baseline to 10 weeks, baseline to 9 months for analysis of effect. The PSS measures the degree to which situations are appraised as stressful. It is a self-report scale with 10 items on daily hassles and the current feeling of being able to handle problems that need to be addressed. It is a five-point Likert scale ranging from 0 (never) to 4 (very often). It is a widely used questionnaire to measure perceived stress and has adequate internal and test-retest reliability.
Pain reactivity Scale (PRS) | Baseline to 10 weeks, baseline to 9 months,
  Change in pain reactivity measured with a self-report scale, pain reactivity scale (PRS), at baseline to 10 weeks, baseline to 9 months. PRS have 5 items about reactivity to and worry about pain. Three items are about emotional reactions to current pain. Two items affect frequency of worry about not being able to do things now, and in the future because of the pain. Questions are answered on a 6-point scale from 0 ("not at all") to 6 ("very much"). PRS has been reported to have satisfactory psychometric properties (Wicksell et al, 2011)
Pain interference index (PII) | Baseline to 10 weeks, baseline to 9 months.
  Change in pain interference measured with a self-report scale at baseline to 10 weeks, baseline to 9 months. Pain interference index (PII), have 6 items about interference on various activities because of pain. Questions are answered on a 6-point scale from 0 ("not at all") to 6 ("very much"). According to preliminary analysis, the instrument has satisfactory psychometric properties (Wicksell et al., 2011)
Functional disability index (FDI) | Baseline to 10 weeks, baseline to 9 months.
  Change in function measured with a self-report scale at baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months. Functional disability index (FDI) have15 items on daily activities. Questions are related to specific activities such as climbing stairs, running 100 meters and to go shopping, and general activities such as eating meals and being in school all day. The scale ranges from 1 (no problem at all) to 5 (impossible). It is validated for children and adolescents with chronic abdominal pain with high internal consistency, α = .86 for boys and α = .91 for girls (Claar and Walker, 2006). FDI is the scale that is recommended in pediatric pain studies to measure the influence of pain on function (McGrath et al., 2008).
Visceral sensitivity Index (IBS-VSI) | Baseline to 10 weeks, baseline to 9 months.
  Change in visceral sensitivity from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures gastrointestinal symptom-specific anxiety. VSI is a 15-item scale and has a scale ranging from 0 (not at all) to 5 (totally agree). The scale has demonstrated excellent reliability as well as good content, convergent, divergent and predictive validity.
Pediatric Quality of Life Inventory (PedsQL) Generic Core scales age 13-18 | Baseline to 10 weeks, baseline to 9 months.
  Change in quality of life from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures quality of life in adolescents. PedsQL Generic Core scales is a 23-item scale ranging from 0 (never) to 4 (almost always). The PedsQL is shown to distinguishe between healthy children and adolescents and pediatric patients with acute or chronic health conditions and demonstrate acceptable reliability and validity.
Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptom Scale | Baseline to 10 weeks, baseline to 9 months.
  Change in gastrointestinal symptoms from baseline to 10 weeks, baseline to 9 months, measured with a self-report scale that measures gastrointestinal symptoms in children and adolescents. The PedsQL Gastro is a 9-item scale ranging from 0 (never) to 4 (almost always).
Children´s Somatization Inventory (CSI-24) | Baseline to 10 weeks, baseline to 9 months.
  Change in inner symptoms from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures inner symptoms (e.g., headache, nausea, heart racing) that often, but not necessarily, occur in the absence of identified disease, in children and adolescents. CSI-24 is a 24-item scale ranging from ranging from 0 '(not at all) to 4 (a whole lot).
Spence Children's Anxiety Scale (SCAS-C) | Baseline to 10 weeks, baseline to 9 months.
  Change in anxiety symptoms from baseline to 10 weeks, baseline to 9 months with a self-report scale that measures anxiety symptoms in children and adolescents. SCAS-C is a 45 -item scale ranging from ranging from 0 (never) to 3 (always). SCAS-C has demonstrated high internal consistency, high concurrent validity with other measures of child and adolescent anxiety, and adequate test-retest reliability.
TiC-P Adolescents revised version | Baseline to 10 weeks, baseline to 9 months.
  Change in healthcare utilization and productivity loss from baseline to 10 weeks, baseline to 9 months, measured with a self-report scale that measures healthcare utilization and productivity. The scale has been revised to fit adolescents and consists in our study of 3 items assessing school absenteeism and 6 items assessing healthcare utilization.
TIC-P Parent report | Baseline to 10 weeks, baseline to 9 months
  Change in parents healthcare utilization and productivity loss from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures healthcare utilization and productivity. TIC-P consists of 10 items.
Generalized Anxiety Disorder Screener (GAD-7) | Baseline to 10 weeks, baseline to 9 months
  Change in anxiety levels in parents from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures anxiety symptoms. GAD-7 is a 7-item scale ranging from 0 (not at all) to 3 (almost every day). Evidence supports reliability and validity of the GAD-7 as a measure of anxiety in the general population.
Patient Health Questionnaire (PHQ 9) | Baseline to 10 weeks, baseline to 9 months
  Change in depression levels in parents from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures depression. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). PHQ-9 is shown to be a reliable and valid measure of depression severity in adults.
ARCS | Baseline to 10 weeks, baseline to 9 months
  Change in parents responses to their children's abdominal pain from baseline to 10 weeks, baseline to 9 months measured with a self-report scale assessing protectiveness, minimizing, and encouraging responses to children's pain behavior. The ARCS is a 29-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Brjánn Ljótsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- BUP-CPF, CAP Research Center, Stockholm, Stockholms County, Sweden

IPD SHARING:
Plan to Share IPD: No